CLINICAL TRIAL: NCT07295678
Title: Open-label Clinical Investigation to Evaluate the Performance and Safety of Medical Device "Urgo Filmocream Eczema" in Association With Dermocorticoids on Atopic Dermatitis Lesions
Brief Title: URGO FilmoCream Eczema + Dermocorticoids in Atopic Dermatitis
Acronym: GERONIMO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CEN Biotech (Industry)
Collaborators: Eurofins Dermscan Pharmascan (Industry); URGO Recherche, Innovation et Développement (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22E4474
Record Dates: First submitted 2025-11-25; First posted 2025-12-19 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Atopic Dermatitis
Keywords: eczema lesions; adjuvant treatment to dermocorticoids; URGO FilmoCream Eczema
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Intervention Model Description: In this intra-individual randomized design, each subject will have two comparable AD lesions, each randomized to receive either URGO FilmoCream Eczema + Desonide 0.1% cream or Desonide 0.1% cream alone.
Who Masked: Outcomes Assessor
Masking Description: Evaluation of the lesions is carried out by a blind observer who is unaware of the treatment allocation of the lesions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- URGO FilmoCream Eczema plus dermocorticoid (Experimental): During the treatment period, URGO FilmoCream Eczema is used alone in the morning and in combination with a topical corticosteroid in the evening.
  During the follow-up phase, it is applied only in case of relapse, twice daily. If the lesion does not improve or worsens, it must be combined with a dermocorticoid in the evening, as during the treatment period.
  Interventions: Combination Product: Treatment period with combination of URGO FilmoCream Eczema and dermocorticoid; Combination Product: Follow-up period after treatment with URGO Filmocream Eczema associated with dermocorticoid
- Dermocorticoid alone (Active Comparator): During the treatment period, a dermocorticoid is used. During the follow-up phase, dermocorticoid is applied only in case of relapse.
  Interventions: Drug: Treatment period with dermocorticoid alone; Drug: Follow-up period after dermocorticoid treatment alone

INTERVENTIONS:
Drug: Treatment period with dermocorticoid alone — Until lesion resolution, for a maximum of 30 consecutive days Treatment with dermocorticoids - desonide 0.1%, or betamethasone 0.05% in case treatment escalation is required.
  Arms: Dermocorticoid alone
Combination Product: Treatment period with combination of URGO FilmoCream Eczema and dermocorticoid — Until lesion resolution, for a maximum of 30 consecutive days URGO FilmoCream Eczema is applied at least twice daily (morning and evening) in a thin layer over the entire surface of the selected lesion, extending 1 cm beyond the edges, and left to dry for about 30 seconds to form a protective film. Reapplication is allowed if the film is disturbed (e.g., due to water exposure), with a maximum of 20 pump pressures per day. In the evening, it is applied after the dermocorticoid - desonide 0.1%, or betamethasone 0.05% in case treatment escalation is required.
  Arms: URGO FilmoCream Eczema plus dermocorticoid
Combination Product: Follow-up period after treatment with URGO Filmocream Eczema associated with dermocorticoid — During the 28-day follow-up period, in case of relapse, URGO FilmoCream Eczema is reapplied twice daily (morning and evening). If there is no improvement or worsening, the combined treatment must be reinitiated under the same conditions as during the treatment period.
  Arms: URGO FilmoCream Eczema plus dermocorticoid
Drug: Follow-up period after dermocorticoid treatment alone — During the 28-day follow-up period, in case of relapse, start with desonide 0.1%, escalate to betamethasone 0.05% if necessary.
  Arms: Dermocorticoid alone

SUMMARY:
The goal of this clinical study is to determine whether URGO FilmoCream Eczema is effective as a non-steroidal treatment to relieve symptoms of atopic dermatitis. It also aims to evaluate the cream's ability to moisturize, soothe irritation, protect the skin, and promote healing of eczema lesions. The main questions the study seeks to answer are:

1. Does URGO FilmoCream Eczema improve symptom relief of atopic dermatitis when used alongside standard topical corticosteroid treatment?
2. How do eczema lesions treated with topical corticosteroids alone progress and heal compared to those treated with topical corticosteroids plus URGO FilmoCream Eczema? To investigate this, patients with at least two similar eczema lesions are enrolled. One lesion is treated with topical corticosteroids alone, while the other is treated with topical corticosteroids plus URGO FilmoCream Eczema.

The progression of both lesions is monitored throughout treatment, until healing, and for 28 days after the last application of topical corticosteroids.

DETAILED DESCRIPTION:
This study has two parts.

1. Treatment phase (up to 30 days):

* For the lesions treated with the combination of both products, URGO FilmoCream Eczema is applied at least twice a day, in the morning and evening. In the evening, it is applied after topical corticosteroid (Desonide 0.1% or, if needed, betamethasone 0.05%).
* For the lesion treated with topical corticosteroid only: treatment starts with Desonide 0.1% and may switch to betamethasone 0.05% if needed.

This part lasts until the skin is fully healed.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject.
2. Aged 18 or more.
3. With mild to moderate atopic dermatitis based on the Investigator's Global Assessment for Atopic Dermatitis (IGA-AD).
4. Presence of two comparable atopic dermatitis lesions requiring treatment with topical corticosteroids, located at anatomically distant sites.
5. Having given her/his informed, written consent,
6. Cooperative, fully informed of the treatment procedures, and aware of the importance and schedule of follow-up visits, ensuring expected full adherence to the study protocol.
7. Psychologically capable of understanding the study information and providing informed consent.
8. Affiliated to a health social security system.
9. Female of childbearing potential should use a contraceptive regimen recognized as effective since at least 12 weeks before screening visit, during all the study and at least 1 month after the study end and must have a negative urine pregnancy test before the first treatment.

Exclusion Criteria:

1. Subject currently participating in another clinical study that may interfere with the assessments of the present study, according to the investigator's judgment.
2. Subject unable to understand the information provided - including study procedures - due to linguistic or psychiatric reasons, and therefore unable to give written informed consent or to complete the study diary as required.
3. Subject who, in the investigator's judgment, is unlikely to comply with study-related constraints and requirements.
4. Subject who has forfeited his/her freedom by administrative or legal decision, or who is under legal guardianship.
5. Female subject of childbearing potential who is pregnant, breastfeeding, or planning to become pregnant during the study.
6. Subject with a known contraindication to topical corticosteroids, such as hypersensitivity to desonide, betamethasone, or any component of the prescribed corticosteroid formulations.
7. Subject with broken or ulcerated skin, acne, rosacea (including perioral dermatitis), any untreated or active skin infection (viral, bacterial, or fungal), or skin thinning at the application sites.
8. Subject with a skin disease, abnormality, or dermatological condition in the study area that may interfere with study assessments.
9. Subject with acute, chronic, or progressive disease, or relevant medical history, considered by the investigator to be hazardous for the subject, incompatible with the study, or likely to interfere with study assessments.
10. Any systemic treatment, including oral corticosteroids, that is incompatible with the study or likely to interfere with study assessments according to the investigator, administered in the weeks prior to the inclusion visit, ongoing, or planned to start during the study.
11. Any topical treatment on the tested area that is incompatible with the study or likely to interfere with study assessments according to the investigator, administered in the weeks prior to the inclusion visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in local SCORAD Index at end of treatment | up to 30 days
  The local SCORAD Index includes the intensity part of SCORAD (SCORing Atopic Dermatitis) index which consists of six signs-erythema, edema/papulation, oozing/crusting, excoriation, lichenification, and xerosis-each rated from 0 (absent) to 3 (severe). The total score is the sum of the 6 items and ranges from 0 to 18, with higher scores indicating more severe local inflammation.
  The variations from baseline in the Local SCORAD Index are compared between lesions treated with the combination therapy and lesions treated with dermocorticoid alone.
Change from baseline in local SCORAD Index at 3 days | 3 days
  The variations from baseline at 3 days in the Local SCORAD (SCORing Atopic Dermatitis) Index are compared between lesions treated with the combination therapy and those treated with dermocorticoid alone. The local SCORAD Index includes the intensity part of SCORAD index which consists of six signs-erythema, edema/papulation, oozing/crusting, excoriation, lichenification, and xerosis-each rated from 0 (absent) to 3 (severe). The total score is the sum of the 6 items and ranges from 0 to 18, with higher scores indicating more severe local inflammation.
Change from baseline in local SCORAD Index at 7 days | 7 days
  The variations from baseline at 7 days in the Local SCORAD (SCORing Atopic Dermatitis) Index are compared between lesions treated with the combination therapy and those treated with dermocorticoid alone. The local SCORAD Index includes the intensity part of SCORAD index which consists of six signs-erythema, edema/papulation, oozing/crusting, excoriation, lichenification, and xerosis-each rated from 0 (absent) to 3 (severe). The total score is the sum of the 6 items and ranges from 0 to 18, with higher scores indicating more severe local inflammation.

SECONDARY OUTCOMES:
Change from baseline in pruritus severity at 3 days | 3 days
  Severity is assessed using a visual analog scale (0-10 VAS), where 0 means no itch and 10 the worst imaginable itch.
  The variations from baseline in 0-10 VAS values are compared between lesions treated with the combination therapy and lesions treated with dermocorticoid alone.
Change from baseline in pruritus severity at 7 days | 7 days
  Severity is assessed using a visual analog scale (0-10 VAS), where 0 means no itch and 10 the worst imaginable itch.
  The variations from baseline in 0-10 VAS values are compared between lesions treated with the combination therapy and lesions treated with dermocorticoid alone.
Change from baseline in pruritus severity at end of treatment | up to 30 days
  Severity is assessed using a visual analog scale (0-10 VAS), where 0 means no itch and 10 the worst imaginable itch.
  The variations from baseline in 0-10 VAS values are compared between lesions treated with the combination therapy and lesions treated with dermocorticoid alone.
Time to complete lesion resolution | 30 days
  Complete resolution is subjectively assessed by the investigator. The time to complete resolution is compared between the two lesion treatments using Kaplan-Meier survival analysis, with differences assessed by the log-rank test.
Dermocorticoid use during the treatment period | 30 days
  The average number of applications of desonide 0.1% and Betamethasone 0.05% will be compared between lesions treated with combination therapy and those treated with dermocorticoid alone.
Relapse rate after initial treatment | 28 days
  Proportions of lesions that relapse after having achieved resolution during the treatment period are compared between lesions treated with the combination therapy and lesions treated with dermocorticoid alone.
Time to the first relapse after initial treatment | 28 days
  The time to the first relapse after initial treatment is compared between the two lesion treatments using Kaplan-Meier survival analysis, with differences assessed by the log-rank test
Dermocorticoid use in relapsed lesions | 28 days
  The average number of applications of desonide 0.1% and Betamethasone 0.05% will be compared between relapsed lesions initially treated with the combination therapy and those initially treated with dermocorticoid alone.

OTHER OUTCOMES:
Change in skin hydration at 3 days | 3 days
  Skin hydration is assessed using the Corneometer® CM 825 (COURAGE & KHAZAKA), which measures the electrical capacitance of the skin surface. This parameter reflects the moisture level of the skin, providing an estimate of its hydration status. The results (hydration index) are expressed in arbitrary units (a.u.).
  The variations from baseline in hydration index values are compared between lesions treated with the combination therapy and lesions treated with dermocorticoid alone.
Change in skin hydration at 7 days | 7 days
  Skin hydration is assessed using the Corneometer® CM 825 (COURAGE & KHAZAKA), which measures the electrical capacitance of the skin surface. This parameter reflects the moisture level of the skin, providing an estimate of its hydration status. The results (hydration index) are expressed in arbitrary units (a.u.).
  The variations from baseline in hydration index values are compared between lesions treated with the combination therapy and lesions treated with dermocorticoid alone.
Change in skin hydration at the end of the treatment | up to 30 days
  Skin hydration is assessed using the Corneometer® CM 825 (COURAGE & KHAZAKA), which measures the electrical capacitance of the skin surface. This parameter reflects the moisture level of the skin, providing an estimate of its hydration status. The results (hydration index) are expressed in arbitrary units (a.u.).
  The variations from baseline in hydration index values are compared between lesions treated with the combination therapy and lesions treated with dermocorticoid alone.
Change in skin barrier integrity at 3 days | 3 days
  Transepidermal Water Loss (TEWL) is measured using a Tewameter TM 300®. And expressed in grams per hour per square meter (g/h/m²). It quantifies the amount of water evaporating from the skin surface over one hour per unit area, providing an indicator of skin barrier function.
  The variations from baseline in TEWL values are compared between lesions treated with combination therapy and lesions treated with dermocorticoid alone.
Change in skin barrier integrity at 7 days | 7 days
  Transepidermal Water Loss (TEWL) is measured using a Tewameter TM 300®. And expressed in grams per hour per square meter (g/h/m²). It quantifies the amount of water evaporating from the skin surface over one hour per unit area, providing an indicator of skin barrier function.
  The variations from baseline in TEWL values are compared between lesions treated with combination therapy and lesions treated with dermocorticoid alone.
Change in skin barrier integrity at the end of the treatment | up to 30 days
  Transepidermal Water Loss (TEWL) is measured using a Tewameter TM 300®. And expressed in grams per hour per square meter (g/h/m²). It quantifies the amount of water evaporating from the skin surface over one hour per unit area, providing an indicator of skin barrier function.
  The variations from baseline in TEWL values are compared between lesions treated with combination therapy and lesions treated with dermocorticoid alone.
Local tolerance to the treatments at Day 3 | 3 days
  Based on patient's reported clinical signs (pain, burning sensation, itching, discomfort or other symptoms) following application of the assigned treatment to the lesion, the investigator subjectively assesses tolerance using a 0-3 scale where 0= Poor tolerance at application, 1= Moderate tolerance at application, 2= Good tolerance at application, 3= Very good tolerance at application.
  Scores are compared between lesions treated with the combination therapy and lesions treated with dermocorticoid alone.
Local tolerance to the treatments at Day 7 | 7 days
  Based on patient's reported clinical signs (pain, burning sensation, itching, discomfort or other symptoms) following application of the assigned treatment to the lesion, the investigator subjectively assesses tolerance using a 0-3 scale where 0= Poor tolerance at application, 1= Moderate tolerance at application, 2= Good tolerance at application, 3= Very good tolerance at application.
  Scores are compared between lesions treated with the combination therapy and lesions treated with dermocorticoid alone.
Local tolerance to the treatments at the end of the treatment | up to 28 days
  Based on patient's reported clinical signs (pain, burning sensation, itching, discomfort or other symptoms) following application of the assigned treatment to the lesion, the investigator subjectively assesses tolerance using a 0-3 scale where 0= Poor tolerance at application, 1= Moderate tolerance at application, 2= Good tolerance at application, 3= Very good tolerance at application.
  Scores are compared between lesions treated with the combination therapy and lesions treated with dermocorticoid alone.
Occurrence of adverse events during the study | up to 58 days
  Adverse events are described using MedDRA , whether they occur during the treatment period or during the follow-up period. Where appropriate, the frequency of treatment adverse effects is compared between lesions treated with the combination therapy and lesions treated with dermocorticoid alone.

CONTACTS AND LOCATIONS:
Overall Officials: Ewa Karamon, Principal Investigator
Locations (2):
- Poland (2):
  - Eurofins Dermscan Poland, Gdansk
  - Private Practice, Malbork

IPD SHARING:
Plan to Share IPD: No
Patient data is not anonymized. To comply with European regulations, patients are informed that no sharing of IPD is planned in order to protect their personal data. Only aggregated data can be shared.